CLINICAL TRIAL: NCT03831243
Title: A Phase III Randomized-controlled, Single-blind Trial to Improve Quality of Life With Stereotactic Body Radiotherapy for Patients With Painful Bone Metastases
Brief Title: A Trial to Improve Quality of Life With Stereotactic Body Radiotherapy for Patients With Painful Bone Metastases
Acronym: ROBOMET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Research Antwerp (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CTOR18072GZA
Record Dates: First submitted 2018-10-22; First posted 2019-02-05 (Actual); Last update posted 2024-02-07 (Actual); Status verified 2022-03

CONDITIONS: Metastasis to Bone; Radiotherapy; Neoplasm Metastasis
Keywords: Stereotactic Body Radiotherapy; Spinal metastases; Bone metastases
MeSH Terms: conditions — Neoplasm Metastasis | interventions — Radiosurgery

STUDY DESIGN:
Intervention Model Description: All subjects will be randomly assigned in a 1:1 ratio to receive either a single fraction of 8.0 Gy to the painful bone metastasis through 3D-CRT (control arm) or a single fraction of 20.0 Gy to the painful bone metastasis through SBRT (experimental arm).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single fraction of 8 Gy (Active Comparator): The current standard treatment will be prescribed, i.e. a 3D-conformal radiotherapy of a single fraction dose of 8.0 Gy to the metastasis with a planning target volume (PTV) margin for set-up and positioning uncertainties of 1 cm. This can be performed at any linear accelerator.
  Interventions: Radiation: 3D-conformal radiotherapy
- Single fraction of 20 Gy (Experimental): Within the framework of stereotactic body radiotherapy, a single fraction dose of 20.0 Gy will be delivered to the metastasis using a PTV margin of 3-5 mm based on high-precision image-guided radiotherapy (IGRT). Therefore, only linear accelerators with the European Organization for Radiotherapy & Oncology advisory committee on radiation oncology practice (ESTRO-ACROP) specifications for SBRT can be accepted. A risk-adapted approach will be applied, aiming for the highest possible dose no less than 16 Gy, while respecting the tolerances of critical organs at risk (e.g. spinal cord, cauda equina, brainstem etc.).
  Interventions: Radiation: Stereotactic body radiotherapy

INTERVENTIONS:
Radiation: Stereotactic body radiotherapy — Treatment will be prescribed to the periphery of the target, i.e. 80% of the dose should cover 95% of the PTV. The organ at risk (OAR) dose constraints will be in accordance with the recommendations from the report of the American Association of Physicists in Medicine (AAPM) task group 101. Image-guidance will consist of cone-beam CT in combination with 6 degrees of freedom corrections using robotic couch.
  Arms: Single fraction of 20 Gy
Radiation: 3D-conformal radiotherapy — In the standard setting, 95% of the PTV should receive 95% of the prescribed dose while near maximum dose (Dnear-max) in the PTV should not exceed 107%. Image-guidance will consist of portal images showing the relevant bony anatomy.
  Arms: Single fraction of 8 Gy

SUMMARY:
This is a phase III randomized-controlled, single-blind study comparing the standard schedule for antalgic radiotherapy of a single fraction of 8.0 Gy delivered through three-dimensional conformal radiotherapy (3D-CRT) to a single fraction of 20.0 Gy delivered through stereotactic body radiotherapy (SBRT). The primary aim of this trial is to double the complete response rate. Secondary aims are to compare general response rates, duration of pain response, acute and late toxicity, HRQoL through patient-reported outcome measures (PROMs), pain flare, and re-irradiation need.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed malignancy.
* Pain score ≥ 2 on a scale from 0 to 10.
* Radiological or (bone) scintigraphic evidence of bone metastasis at the site of pain.
* Lesions ≤ 5cm in largest diameter.
* Per lesion no more than 3 consecutive spine segments involved with one unaffected vertebral body above and below.
* No more than 3 painful lesions needing treatment.
* Life expectancy estimated at > 3 months.
* Patients who have received the information sheet and signed the informed consent form.
* Patients must be willing to comply with scheduled visits, treatment plan, and other study procedures.
* Patients with a public and/or private health insurance coverage.

Exclusion Criteria:

* Myeloma.
* Bone metastasis in previously irradiated sites.
* Previous radioisotope treatment for bone metastases.
* Complicated bone metastasis, i.e. impending and/or existing pathological fracture, spinal cord compression or cauda equina compression [16].
* Patients with significantly altered mental status or with psychological, familial, sociological or geographical condition potential hampering compliance with the study.
* Individual deprived of liberty or placed under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2019-04-09 (Actual); Primary Completion 2023-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
Pain response | 4 weeks after RT visit
  Pain response at the treated index site at 1 month after radiotherapy (RT), as defined by the consensus statement.

SECONDARY OUTCOMES:
Incidence of pain flare | 24-48 hours after radiotherapy
  Number of participants with increase in pain score of 2 or more above baseline at the treated site with stable OMED, or an increase of 25% or more in OMED compared with baseline with the pain score stable or 1 point above baseline
Duration of pain response | 2 years after radiotherapy
  Time until pain progression (defined as an increase in pain score of 2 or more above baseline at the treated site with stable daily oral morphine equivalent, or an increase of 25% or more in daily oral morphine equivalent (OMED) compared with baseline with the pain score stable or 1 point above baseline)
Re-irradiation need | 2 years after radiotherapy
  Need for re-irradiation of the treated lesion
Acute toxicity Measured with CTCAE version 5.0 | 3 months after radiotherapy
  Measured with CTCAE version 5.0
Late toxicity Measured with CTCAE version 5.0 | 2 years after radiotherapy
  Measured with CTCAE version 5.0
Impact of treatment on Quality of Life: EORTC quality of life questionnaire (QLQ) BM22 | 2 years after radiotherapy
  Using the EORTC quality of life questionnaire for Bone Metastases (QLQ BM22) to measure impact of bone metastases on QoL [min score 0 - max score 100]. A high score represents a high level of symptomatology. The score is calculated by applying a linear transformation on the scores to each answer of the 22 question-long questionnaire (cfr. EORTC mannual).
Number of Subsequent Serious Skeletal events | 2 years after radiotherapy
  Incidence of symptomatic pathologic fractures, radiation or surgery to bone, and spinal cord compression.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Verellen, PhD, Study Director — Iridium Cancer Network
Locations (1):
- Radiotherapy department, GZA Hospitals, Wilrijk, Antwerp, Belgium

REFERENCES:
- [Derived] Mercier C, Billiet C, Ost P, Vandecasteele K, De Kerf G, Claessens M, Van Laere S, Vermeulen P, Dirix L, Lievens Y, Verellen D, Dirix P. Dose-Escalated Stereotactic Versus Conventional Radiotherapy for Painful Bone Metastases (ROBOMET): A Multicenter, Patient-Blinded Randomized Clinical Trial. J Clin Oncol. 2025 Jul;43(19):2164-2172. doi: 10.1200/JCO-24-01447. Epub 2025 May 8. PMID 40340551
- [Derived] Mercier C, Dirix P, Ost P, Billiet C, Joye I, Vermeulen P, Lievens Y, Verellen D. A phase III randomized-controlled, single-blind trial to improve quality of life with stereotactic body radiotherapy for patients with painful bone metastases (ROBOMET). BMC Cancer. 2019 Sep 4;19(1):876. doi: 10.1186/s12885-019-6097-z. PMID 31484505